CLINICAL TRIAL: NCT04357080
Title: Factors Predicting Urethral Stricture Recurrence After Dorsal Onlay Augmented, Buccal Mucosal Graft Urethroplasty
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor of Urology and Andrology, Al-Azhar University
Other Study IDs: Uro_Azhar_4_020
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-04

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with urethral stricture recurrence
  Interventions: Procedure: Urethroplasty
- Control: Patients with normal, patent urethra
  Interventions: Procedure: Urethroplasty

INTERVENTIONS:
Procedure: Urethroplasty — Augmentation Anterior Urethroplasty Using Dorsal Onlay Buccal Mucosal Graft

SUMMARY:
In this observational study, the investigators will evaluate potential risk factors associated with urethral stricture recurrence after augmentation anterior urethroplasty using dorsal onlay buccal mucosal Graft during the past 10 years. Patients' medical files will be reviewed for data relevant to demographics, clinical and operative characteristics. data will be analyzed using the appropriate statistical tests and the independent predictors of urethroplasty outcome will be identified.

DETAILED DESCRIPTION:
In this series, the investigators will study different factors related to the stricture and to the patients to identify the independent predictors of urethral stricture recurrence after augmentation anterior urethroplasty using dorsal onlay buccal mucosal graft.

A retrospective review of medical records will be performed to identify patients who underwent augmented anastomotic anterior urethroplasty with dorsal onlay graft at Al-Azhar University Hospitals in Egypt since 2010. Patients will be included only if they were two or more years out of surgery. The data will be recorded without patients' identification.

Data to be collected are patient age, body mass index (BMI), smoking status, diabetes status, overall comorbidity, stricture etiology, prior endoscopic treatment and open urethroplasty, urethral stricture length and location, degree of urethral obliteration, urethral plate width, presence and degree of spongiofibrosis. estimated intraoperative blood loss, catheter size, overall operative time, hospital stay and early postoperative complications.

The diagnosis of urethral stricture recurrence is based on the radiological and endoscopic features of stricture recurrence. Time to recurrence will be calculated from the date of surgery till the date restricture diagnosis.

Univariate and multivariate regression analysis will be performed and factors predicting urethral stricture recurrence will be identified.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be 2 years or more out of surgery

Exclusion Criteria:

* patients with incomplete medical records or follow-up informations

Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male of any age
Study Population: patients who underwent augmented anterior urethroplasty with buccal mucosal graft at Al-Azhar University Hospital in the past 10 years
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
urethral restricture rate | At any time from date of surgery until the last follow-up visit (up to 10 years)
  The presence of radiologic and endoscopic features of urethral stricture recurrence, as diagnosed by urethrography and cystoscopy during follow-up.
Time to urethral restricture. | The time from urethroplasty surgery until the time of urethral restricure diagnosis (at any follow-up time point, up to 10 years), as recorded in patients medical files).
  will be calculated from the date of surgery until the date restricture diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided